CLINICAL TRIAL: NCT06909825
Title: A Phase 2, Open-label, Multi-centre Study of FPI-2265 (225Ac-PSMA-I&T) and Olaparib in Participants With Metastatic Castration Resistant Prostate Cancer (mCRPC)
Brief Title: FPI-2265 (225Ac-PSMA-I&T) and Olaparib for Patients With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fusion Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FPI-2265-203; CT-2024-CTN-00137-1 (Other: TGA Clinical Trial Notification (CTN))
Record Dates: First submitted 2025-03-21; First posted 2025-04-04 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: mCRPC; 225Ac-PSMA-I&T; RLT; Radioligand Therapy; FPI-2265; Olaparib; Radioconjugate
MeSH Terms: interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part A (Experimental): Regimen 1: FPI-2265 (Dose A intravenously [IV] every six weeks) plus olaparib (twice daily [BID], on Days 1 to 14 of each cycle).
  Regimen 2: . FPI-2265 (Dose B intravenously [IV] every 4 weeks) plus olaparib (twice daily [BID], on Days 1 to 14 of each cycle)
  Interventions: Drug: FPI-2265; Drug: Olaparib
- Part B (Experimental): Regimen 1: FPI-2265 (Dose A intravenously [IV] every six weeks) plus olaparib (g twice daily [BID], on Days 1 to 14 of each cycle).
  Regimen 2: . FPI-2265 (Dose B intravenously [IV] every 4 weeks) plus olaparib (twice daily [BID], on Days 1 to 14 of each cycle)
  Interventions: Drug: FPI-2265; Drug: Olaparib

INTERVENTIONS:
Drug: FPI-2265 — PSMA ligand radiolabeled with Ac225
Drug: Olaparib — Poly (ADP-ribose) polymerase (PARP) inhibitor

SUMMARY:
This study is an open-label, multicenter study designed to investigate the efficacy, safety and tolerability of FPI-2265 (225Ac-PSMA-I&T) in combination with Olaparib in participants with mCRPC. The dose optimization Phase 2 part will be investigating the safety, tolerability, and anti-tumor activity of novel dosing regimens of FPI-2265 and Olaparib in participants with metastatic castration-resistant prostate cancer.

DETAILED DESCRIPTION:
This study is an open-label, multicenter study designed to investigate the efficacy, safety and tolerability of FPI-2265 (225Ac-PSMA-I&T) in combination with Olaparib in participants with mCRPC. The study will be conducted in two parts, with Part A enrolling participants who have been previously treated with lutetium-177 (177Lu) vipivotide tetraxetan or other 177Lu-PSMA radioligand therapy (RLT) and Part B enrolling participants who have not been previously treated with lutetium-177 (177Lu) vipivotide tetraxetan or other 177Lu-PSMA radioligand therapy. For each part of the study, a Simon 2-stage design will be used to evaluate two dosing regimens. The purpose of this investigation is to determine the recommended FPI-2265 dose and regimen. Conclusions from this Phase 2 study will be based on safety, tolerability, and anti-tumor activity data. Participants with PSMA-positive mCRPC will be allocated to Arm 1 and Arm 2 in a singular, alternating fashion, until all Stage 1 participants are enrolled into each of the two regimens:

Arm 1: Will consist of up to six doses of FPI-2265 every six weeks at Dose A and olaparib twice a day on days 1 to 14 of each cycle.

Arm 2: Will consist of up to nine doses of FPI-2265 every four weeks at Dose B and olaparib twice a day on days 1 to 14 of each cycle Participants will be monitored and assessed for efficacy response, disease progression, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male participants with mCRPC that is progressing at the time of study entry
2. ECOG performance status 0-1 and life expectancy of at least three months
3. Must have received at least one novel anti-androgen deprivation therapy
4. Participants with known BRCA mutations should have received approved therapies such as PARP inhibitors, per Investigator discretion.
5. All prior treatment-related AEs must have resolved to CTCAE Grade ≤1 (except alopecia).
6. Participants must have had prior orchiectomy and/or ongoing androgen deprivation therapy and a castrate level of serum testosterone (<50 ng/dL or <1.7 nmol/L)
7. Positive PSMA PET/CT scans .
8. Participants must have adequate organ and bone marrow function:

   * Hgb >/= 9g/dL
   * Platelets >/= 100 x 10^9/L
   * ANC </= 1.5 x 10^9/L
   * CrCL >/= 50 mL/min

Exclusion Criteria:

1. Previous treatment with any of the following within 6 months of first dose: Samarium-153, Rhenium-186, Rhenium-188, Radium-223, hemi-body irradiation.
2. Participants who received more than two (2) prior lines of cytotoxic chemotherapy for CRPC.
3. Participants with known unresolved urinary tract obstruction.
4. Transfusion- or growth factor-dependent participants.
5. Participants with a history of CNS metastases are excluded, except those who have received therapy (and are neurologically stable, asymptomatic, and not receiving corticosteroids for the purposes of maintaining neurologic integrity.
6. Symptomatic cord compression, or clinical or radiologic findings indicative of impending cord compression.
7. Participants with any liver metastases.
8. Participants with skeletal metastases presenting as a superscan .
9. Previous history of interstitial lung disease or non-infectious pneumonitis.
10. Participants with a history or clinical and/or laboratory features suggestive of MDS/AML.
11. Major surgery ≤28 days prior to the first dose of study treatment.
12. Planning to conceive a pregnancy during the treatment and up to six months after the last treatment.
13. Participants unable to swallow orally administered medications or with malabsorptive gastrointestinal disorders.
14. Concomitant use of known strong or moderate CYP3A inhibitors or inducers

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 85 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2030-01-29 (Estimated); Study Completion 2030-08-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate anti-tumour activity of FPI-2265 administered in combination with olaparib | From first dose until approximately 12 weeks after the first administered dose of FPI-2265
  The frequency and proportion of participants with PSA50 response will be summarized, where PSA50 is defined as ≥50% decline in PSA level from pre-treatment.
Evaluate the safety and tolerability of FPI-2265 administered in combination with olaparib | From first dose until end of long-term follow-up, 5 years from the last administered dose of FPI-2265
  Safety will be assessed by percentage of patient with treatment emergent adverse events and serious adverse events; percentage of patients with SAEs during the first year of the long term follow up and the number of AESIs during the 5 year follow up period. Percentage of patients with interruption of FPI-2265; percentage of patients who discontinue treatment; number and grade for AEs related to study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dipti Shoop, Study Director — Fusion Pharmaceuticals Inc.
Locations (4):
- Australia (4):
  - Macquarie University Hospital, Macquarie Park, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Icon Cancer Centre Kurralta Park, Kurralta Park, South Australia
  - Peter MacCallum Cancer Center, Melbourne, Victoria